CLINICAL TRIAL: NCT04330469
Title: Effect of Periodontal Therapy and Modification of Oral-gut-hepatic Axis in Patients With Cirrhosis
Brief Title: Periodontal Therapy and Oral-gut-hepatic Axis Cirrhosis: a Randomized Controlled Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Madhumita Premkumar, Assistant professor, Department of heaptology, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IEC/11/2019/1396
Record Dates: First submitted 2020-03-23; First posted 2020-04-01 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Periodontal Diseases; Cirrhosis
Keywords: Periodontitis; Cirrhosis
MeSH Terms: conditions — Periodontal Diseases; Fibrosis; Periodontitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Periodontal therapy (Experimental): Patients offered periodontal therapy in 2-4 sittings (n=40), Dental hygiene advised
  Interventions: Procedure: Periodontal therapy
- Control (Sham Comparator): Patients given standard medical treatment (n=40), Dental hygiene advised
  Interventions: Procedure: Oral hygiene advice

INTERVENTIONS:
Procedure: Periodontal therapy — Treatment will be performed by a periodontist.
  1. Intensive removal of subgingival and supragingival calculus and plaque biofilm by scaling, root-planing and polishing. The procedures will be carried out with the use of hand scalers and a piezoelectric ultrasonic scaler with universal tips. Disclosing solution will be used to visualize the plaque for the clinician.
  2. One to four sessions of subgingival scaling and root planing by quadrant, under local anesthesia as may be deemed necessary during the study period.
  3. Subgingival irrigation using an antiseptic mouth rinse (chlorhexidine 0.12%).
  4. Polishing of the coronal and radicular surfaces of the teeth.
  Arms: Periodontal therapy
Procedure: Oral hygiene advice — Oral hygiene advised by Periodontist
  Arms: Control

SUMMARY:
Periodontitis is common in patients with cirrhosis and may lead to systemic sepsis. 1 Grønkjær et al demonstrated that severe periodontitis predicted higher mortality in patients with cirrhosis. 2 In India, the wide use of oral tobacco, smoking and poor dental hygiene fosters a dual hit to the outcomes of liver disease especially in the setting of liver transplantation. However, a causal relationship between the oral microbiome and liver disease and outcomes is a matter of conjecture. Oral bacterial diseases, such as caries and periodontitis are caused by a consortium of bacteria rather than a single species. These constitute opportunistic infections that occur under the proper circumstances and conditions, e.g., diet, host immune response, complicating systemic or genetic disorders, pH, poor oral hygiene and lifestyle. It is well known that specific bacterial taxa that colonize the oral cavity are associated with oral health and oral diseases or afflictions, such as dental caries, periodontal diseases, endodontic lesions, dry socket, halitosis, and odontogenic infections.

Bajaj et al have demonstrated systematic periodontal therapy in cirrhotic outpatients improved endotoxemia, as well as systemic and local inflammation, and modulated salivary and stool microbial dysbiosis over 30 days. Bajaj et al performed another study on comparison of oral and gut microbiota in patients with and without hepatic encephalopathy.

There were differences in salivary microbiota composition and inflammatory markers between controls and cirrhotics. The association between periodontitis, oral dysbiosis and the prognosis of cirrhosis remains crucial with relevance to situations like acute-on-chronic liver failure and other inflammation-related adverse events.

DETAILED DESCRIPTION:
The aim of this study is to prospectively determine the association of generalised Stage I & II (initial to moderate) with all-cause and cirrhosis-related mortality in patients with cirrhosis. We also plan to evaluate the oral microbiome and association of oral dysbiosis with complications of cirrhosis to assess if early treatment by dental interventions may improve nutrition and outcomes in cirrhosis. Lastly this prospective randomized controlled trial will provide insight into whether manipulation of the oral microbiome by dental procedures and oral hygiene training, antibiotics- local and systemic, use of probiotics etc can alter adverse outcomes, nutrition and health related quality of life in cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

* Cirrhosis of any etiology
* Aged between 18 Years to 65 Years
* Either gender
* Generalized Stage I & II Periodontitis as defined by the 2017 World Workshop on the Classification of Periodontal and Peri-Implant Diseases and Conditions)

Exclusion Criteria:

* Inability to obtain informed consent from patient or relatives.
* Severe cardiopulmonary disease
* Pregnancy
* HIV infection
* Recent abdominal surgery (with in last 6 months)
* Patient on immunosuppressive drugs
* Malignancies including Hepatocellular carcinoma
* Gastrointestinal (GI bleed) in the last 4 weeks
* Oral antibiotics or antifungals taken in last 2 weeks.
* Active sepsis
* Stage III & IV Periodontitis
* Localized /Molar-incisor pattern
* Patients who received periodontal treatment within the last 6 months
* Patients who require antibiotic prophylaxis before examination or treatment
* Presence of a carious exposed teeth/periapical abscess etc requiring Root Canal Treatment/extraction

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-03-01 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
All-cause Hospitalizations | 90days
  All-cause, liver-related and elective hospitalizations at 3 months
Change in Model for End Stage Liver Disease (MELD) score | 90 days

SECONDARY OUTCOMES:
Change in systemic inflammatory cytokines in the blood | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Madhumita Premkumar, DM, Principal Investigator — Post Graduate Institute of Medical Education and Research, Chandigarh
Locations (1):
- Postgraduate Institute of Medical Education and Research, Chandigarh, India

REFERENCES:
- [Background] Costa FO, Lages EJP, Lages EMB, Cota LOM. Periodontitis in individuals with liver cirrhosis: A case-control study. J Clin Periodontol. 2019 Oct;46(10):991-998. doi: 10.1111/jcpe.13172. Epub 2019 Aug 28. PMID 31336404
- [Background] Gronkjaer LL, Holmstrup P, Schou S, Kongstad J, Jepsen P, Vilstrup H. Periodontitis in patients with cirrhosis: a cross-sectional study. BMC Oral Health. 2018 Feb 13;18(1):22. doi: 10.1186/s12903-018-0487-5. PMID 29439734
- [Background] Hanioka T, Morita M, Yamamoto T, Inagaki K, Wang PL, Ito H, Morozumi T, Takeshita T, Suzuki N, Shigeishi H, Sugiyama M, Ohta K, Nagao T, Hanada N, Ojima M, Ogawa H. Smoking and periodontal microorganisms. Jpn Dent Sci Rev. 2019 Nov;55(1):88-94. doi: 10.1016/j.jdsr.2019.03.002. Epub 2019 Apr 24. PMID 31049117
- [Background] Helenius-Hietala J, Meurman JH, Hockerstedt K, Lindqvist C, Isoniemi H. Effect of the aetiology and severity of liver disease on oral health and dental treatment prior to transplantation. Transpl Int. 2012 Feb;25(2):158-65. doi: 10.1111/j.1432-2277.2011.01381.x. Epub 2011 Nov 5. PMID 22054477
- [Background] Aberg F, Helenius-Hietala J, Meurman J, Isoniemi H. Association between dental infections and the clinical course of chronic liver disease. Hepatol Res. 2014 Mar;44(3):349-53. doi: 10.1111/hepr.12126. Epub 2013 Apr 29. PMID 23607641
- [Background] Krishnan K, Chen T, Paster BJ. A practical guide to the oral microbiome and its relation to health and disease. Oral Dis. 2017 Apr;23(3):276-286. doi: 10.1111/odi.12509. Epub 2016 Jul 4. PMID 27219464
- [Background] Bajaj JS, Matin P, White MB, Fagan A, Deeb JG, Acharya C, Dalmet SS, Sikaroodi M, Gillevet PM, Sahingur SE. Periodontal therapy favorably modulates the oral-gut-hepatic axis in cirrhosis. Am J Physiol Gastrointest Liver Physiol. 2018 Nov 1;315(5):G824-G837. doi: 10.1152/ajpgi.00230.2018. Epub 2018 Aug 17. PMID 30118351